CLINICAL TRIAL: NCT03663712
Title: A Phase I Trial of Talimogene Laherparepvec for the Treatment of Peritoneal Surface Malignancies
Brief Title: Talimogene Laherparepvec for the Treatment of Peritoneal Surface Malignancies
Acronym: TEMPO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dan Blazer III, M.D. (Other)
Responsible Party: Sponsor-Investigator, Dan Blazer III, M.D., Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00086917
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Peritoneal Surface Malignancy
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 4 x 10^6 PFU (Experimental): Dose level 1. Subjects were assigned to receive 4 x 10^6 PFU of talimogene laherparepvec.
  Interventions: Biological: Talimogene Laherparepvec
- 4 x 10^7 PFU (Experimental): Dose level 2. Subjects were assigned to receive 4 x 10^7 PFU of talimogene laherparepvec.
  Interventions: Biological: Talimogene Laherparepvec
- 4 x 10^8 PFU (Experimental): Dose level 3. Subjects were assigned to receive 4 x 10^8 PFU of talimogene laherparepvec.
  Interventions: Biological: Talimogene Laherparepvec

INTERVENTIONS:
Biological: Talimogene Laherparepvec — TVEC is an oncolytic, genetically modified virus designed to reproduce in tumor tissue and stimulate your immune system to attack the tumor cells
  Other Names: (T-VEC)

SUMMARY:
The primary objective of this open-label, Phase I, trial is to evaluate the toxicity profile of intraperitoneal talimogene laherparepvec (TVEC) in patients with peritoneal surface dissemination from gastrointestinal or recurrent, platinum-resistant ovarian tumors. The secondary objectives are to evaluate the pharmacokinetic profile and viral shedding of TVEC by measuring viral load in serum and urine as well as viral load in peritoneal washings.

DETAILED DESCRIPTION:
This is a non-randomized, open-label Phase I trial in patients with Stage IV peritoneal surface dissemination from gastrointestinal or recurrent, platinum-resistant ovarian tumors enrolled at Duke Cancer Institute. All subjects will complete an extensive medical history, baseline physical examination and clinical assessment to ensure subject eligibility requirements within 4 weeks of starting study drug. All eligible patients must have a peritoneal catheter placed at least 2 weeks prior to the initiation of therapy. All patients will receive an initial loading dose of TVEC 4x10^6 Plaque Forming Units (PFU) on Cycle 1 Day 1 to enable the formation of protective antibodies as described in the currently approved treatment protocol for the treatment of cutaneous melanoma. Three weeks after the initial loading dose, patients will receive TVEC at the dose level for the cohort for which they are enrolled every 2 weeks for up to 4 doses. The length of the first cycle is 5 weeks and subsequent cycles are 2 weeks in duration.

The first portion of the study, the Dose Escalation cohort, will evaluate the toxicity profile of TVEC in patients with peritoneal surface dissemination from gastrointestinal or recurrent, platinum-resistant ovarian tumors. Using a standard '3+3' dose escalation design, there are up to three dose levels that may be explored. Dose escalation will be dependent on dose-limiting toxicity (DLT) within the cohorts.

Once the maximum tolerated dose (MTD) has been determined, an additional 6 subjects will be enrolled to the dose expansion cohort. All subjects will receive an initial loading dose of TVEC 4x10^6 PFU on Cycle 1 Day 1. Three weeks after the initial loading dose, patients will receive TVEC at the MTD every 2 weeks for up to 4 doses. The length of the first cycle is 5 weeks and the subsequent cycles are 2 weeks in duration. There are a total of four cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have stage IV peritoneal surface dissemination of gastrointestinal cancer or recurrent ovarian, fallopian tube or primary peritoneal cancer with metastatic disease to the peritoneum that cannot be completely resected at time of abdominal exploration. Please note:

   1. Locoregional extension of peritoneal disease beyond the peritoneal cavity (including but not limited to the pleura and subcutaneous soft tissue) is permitted with PI approval,
   2. Radiographically measurable disease is preferable, but for patients with previously documented gastrointestinal, fallopian tube, ovarian, or primary peritoneal cancer, for whom relevant tumor markers (including but not limited to CEA, CA 19-9 or CA-125) have been useful markers of disease progression and/or response to treatment, an elevated relevant tumor marker (including but not limited to CEA, CA 19-9 or CA-125) above the institutional upper limit of normal could be substituted for radiographic imaging,
   3. Asymptomatic primary tumors are permitted.
2. Subjects must have had at least one prior round of systemic therapy or have refused or be ineligible for standard systemic therapy for their disease type. No prior systemic therapy is required for low grade mucinous cancers.
3. Age ≥ 18 years
4. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2
5. Adequate marrow function as evidenced by:

   1. Absolute neutrophil count (ANC) ≥ 2,000/µL
   2. Platelets ≥ 100,000/µL
   3. Hemoglobin (Hgb) ≥ 9 g/dL
6. Adequate renal function as evidenced by serum creatinine ≤ 1.5 x upper limit of normal (ULN), OR 24-hour creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 x ULN.
7. Adequate hepatic function as evidenced by:

   1. Serum bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for a subject with total bilirubin level > 1.5 x ULN
   2. Aspartate aminotransferase (AST) ≤ 3 x ULN
   3. Alanine aminotransferase (ALT) ≤ 3 x ULN
   4. Alkaline phosphatase ≤ 3 x ULN
8. INR or PT ≤ 1.5 x ULN, unless the subject is receiving anticoagulant therapy, in which case PT and PTT/aPTT must be within therapeutic range of intended use of anticoagulants (and may need to be held per institutional standards for placement of the Bard peritoneal catheter).
9. Patients must be recovered from both acute and late effects of any prior surgery, radiotherapy or other antineoplastic therapy.
10. Patients of reproductive potential (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) at the time of pregnancy test (women of childbearing potential only), during the course of the study and for 90 days after the last dose of study drug, even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of study and for 90 days after the last dose of study drug.
11. Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial.

Exclusion Criteria:

1. Prior chemotherapy, radiotherapy, biological cancer therapy, targeted therapy, or major surgery within 28 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment.
2. Patients who received radiotherapy to more than 25% of their bone marrow.
3. Currently receiving treatment with another investigational device or drug study, or < 30 days since ending treatment with another investigational device or drug study(s). Other investigational procedures while participating in this study are excluded.
4. Known active central nervous system (CNS) metastases. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids >10 mg/day of prednisone or equivalent. The exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
5. Metastatic disease in a site other than the peritoneal surfaces. Note: Locoregional extension of peritoneal disease may be permitted with PI approval.
6. History or evidence of active autoimmune disease that requires systemic treatment (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
7. Evidence of clinically significant immunosuppression such as the following:

   1. Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease.
   2. Concurrent opportunistic infection.
   3. Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses >10mg/day of prednisone or equivalent within 7 days prior to enrollment.
8. History of allogenic organ or hematopoietic transplant.
9. Active herpes simplex virus (HSV) that requires intermittent or chronic systemic anti-herpetic therapy or prior complications of herpetic infection, e.g. herpetic keratitis or encephalitis.
10. Requiring intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use.
11. Prior treatment with talimogene laherparepvec or any other oncolytic virus.
12. Subject has known sensitivity to talimogene laherparepvec or any of its components to be administered during dosing.
13. Prior therapy with tumor vaccine.
14. Receipt of a live vaccine within 28 days prior to enrollment.
15. Known to have acute or chronic active hepatitis B or C infection (active, previously treated, or both).
16. Known history of HIV infection.
17. Active infection or fever ≥ 101.3°F within 3 days of the first scheduled day of protocol treatment.
18. Peripheral neuropathy ≥ Grade 2.
19. Bleeding disorders that would preclude intraperitoneal port placement.
20. Refractory ascites that requires palliative paracentesis more frequently than once a month. Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study or interferes with the interpretation of the results.
21. History of other malignancy within the past 5 years.
22. Female subjects who are pregnant or breast-feeding, or planning to become pregnant during study treatment or through 90 days after the last dose of talimogene laherparepvec.
23. Subjects of childbearing potential who are unwilling to use acceptable method(s) of effective contraception during study treatment and through 90 days after the last dose of talimogene laherparepvec.
24. Sexually active subjects and their partners unwilling to use male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 90 days after treatment with talimogene laherparepvec.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Blazer, MD, Principal Investigator — Duke University; John H Stewart, MD, Study Chair — University of Illinois College of Medicine at Chicago
Locations (3):
- United States (3):
  - University of Illinois College of Medicine at Chicago, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 3 sites (Duke University Medical Center, University of Illinois at Chicago, and Wake Forest Baptist Medical Center).
Pre-assignment Details: 28 subjects signed the consent form. 9 failed screening and were withdrawn from the study. 1 voluntarily withdrew from the study before getting the study drug. 18 of them received the study drug and are considered evaluable subjects.
Groups:
- Dose Level 1: 4 x 10^6 Plaque Forming Units (PFU) of talimogene laherparepvec.
- Dose Level 2: 4 x 10^7 Plaque Forming Units (PFU) of talimogene laherparepvec.
- Dose Level 3: 4 x 10^8 Plaque Forming Units (PFU) of talimogene laherparepvec.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 3 | 4 | 11
Completed | 3 | 4 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1: 4 x 10^6 PFU of talimogene laherparepvec.
- Dose Level 2: 4 x 10^7 PFU of talimogene laherparepvec.
- Dose Level 3: 4 x 10^8 PFU of talimogene laherparepvec.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 3 | 4 | 11 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (4.9) | 56.5 (11.0) | 61.2 (7.2) | 61.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 7 | 10
  Male | 1 | 3 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 11 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 2 | 2
  White | 3 | 3 | 9 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: Number of participants who experienced a dose limiting toxicity (DLT)
Time Frame: from start of treatment until 30-day follow-up visit, up to 14 weeks
Measure: Count of Participants; unit: Participants
Groups:
- TVEC Dose of 4x10^6 PFU (Plaque-forming Units): Dose level 1. Subjects were assigned to receive 4 x 10^6 PFU of talimogene laherparepvec.
- TVEC Dose of 4x10^7 PFU (Plaque-forming Units): Dose level 2. Subjects were assigned to receive 4 x 10^7 PFU of talimogene laherparepvec.
- TVEC Dose of 4x10^8 PFU (Plaque-forming Units): Dose level 3. Subjects were assigned to receive 4 x 10^8 PFU of talimogene laherparepvec.
Arm/Group | TVEC Dose of 4x10^6 PFU (Plaque-forming Units) | TVEC Dose of 4x10^7 PFU (Plaque-forming Units) | TVEC Dose of 4x10^8 PFU (Plaque-forming Units)
Number analyzed (Participants) | 3 | 4 | 11
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of treatment until 30-day follow-up visit, up to 14 weeks
Groups:
- Dose Level 1: 4x10^6 PFU of talimogene laherparepvec.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/4 | 5/11
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/4 | 3/11
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=4) | Dose Level 3 (N=11)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
intraperitoneal port obstruction (Gastrointestinal disorders) | 0 | 1 | 0
failure to thrive (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
peritoneal port infection (Infections and infestations) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=4) | Dose Level 3 (N=11)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 8
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 2 | 1
Fatigue (General disorders) | 1 | 2 | 2
Fever (General disorders) | 0 | 2 | 3
Neutrophil count decreased (Investigations) | 1 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT03663712/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT03663712/ICF_001.pdf